CLINICAL TRIAL: NCT01335061
Title: A Multicenter, Open-label Study To Compare On-demand Treatment To A Prophylaxis Regimen Of Nonacog-alfa (Benefix) In Subjects With Moderately Severe To Severe Hemophilia B (Fix:c</=2%)
Brief Title: Study To Compare On-Demand Treatment To A Prophylaxis Regimen Of BeneFIX In Subjects With Moderately Severe to Severe Hemophilia B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B1821010; 3090A1-3306 (Other: Alias Study Number); 2011-000520-15 (EudraCT Number)
Record Dates: First submitted 2011-03-30; First posted 2011-04-13 (Estimated); Results first posted 2015-05-04 (Estimated); Last update posted 2015-06-08 (Estimated); Status verified 2015-05

CONDITIONS: Hemophilia B
Keywords: Hemophilia B; on-demand; prophylaxis; nonacog alfa; BeneFIX; FIX
MeSH Terms: conditions — Hemophilia B | interventions — Factor IX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BeneFIX (Other)
  Interventions: Biological: Nonacog alfa

INTERVENTIONS:
Biological: Nonacog alfa — Period 1: During on-demand period, dosing at the discretion of investigator.
  Other Names: BeneFIX
Biological: Nonacog alfa — Period 2: During the prophylaxis period, 100 IU/kg once weekly
  Other Names: BeneFIX

SUMMARY:
The purpose of this study will be to determine if a once-weekly prophylaxis regimen of BeneFIX in subjects with moderately severe to severe Hemophilia B is safe and effective.

ELIGIBILITY:
Inclusion Criteria:

* Documented history of moderately-severe to severe hemophilia B (FIX activity </=2%).
* Male subjects, aged 12 years to 65 years.
* Subjects with at least 100 exposure days (EDs) to factor IX products.
* Subjects with a minimum of 12 bleeding episodes, 6 of which must be joint bleeds, in the 12-month period before the Screening visit.

Exclusion Criteria:

* Subjects who have received FIX as a primary or secondary prophylaxis regimen within the last 12 months prior to the Screening visit.
* Subjects who have had major surgery or an orthopedic surgical procedure within the past 3 months prior to Screening visit.
* Subjects for which major surgery or orthopedic surgery is planned within the duration of study participation.
* Subjects with a past history of, or current FIX inhibitor, defined as >ULN (upper limit of normal) of the reporting laboratory.
* Subjects with a known hypersensitivity to any FIX product or hamster protein.

Ages: 12 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (17):
- UMBAL Sveti Georgi, Klinika po hematologia, Plovdiv, Bulgaria
- The Ottawa Hospital, Ottawa, Ontario, Canada
- University Hospital Center Zagreb, Zagreb, Croatia
- Malaysia (2):
  - National Blood Centre, Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan, Pahang
- Mexico (2):
  - Instituto Biomedico de Investigacion A.C., Aguascalientes, Aguascalientes
  - Hospital y Clinica OCA, Monterrey, Nuevo León
- Poland (2):
  - Nzoz Triclinium, Warsaw
  - Klinika Hematologii, Nowotworow Krwi i Transplantacji Szpiku, Wroclaw
- Singapore General Hospital, Singapore, Singapore
- Eulji University Hospital, Daejeon, South Korea
- Turkey (Türkiye) (6):
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali Hematoloji Bilim Dali, Fatih, Istanbul
  - Hacettepe Universitesi Tip Fakultesi Ic Hastaliklari Anabilim Dali Hematoloji Bolumu, Ankara
  - Ege Universitesi Tip Fakultesi, Bornova/Izmir
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Arastirma ve Uygulama Hastanesi Hematoloji Poliklinigi, Gaziantep
  - Erciyes Universitesi Tip Fakultesi, Kayseri
  - Erciyes Universitesi Tip Fakultesi Hastaneleri M. Kemal Dedeman Onkoloji Hastanesi, Kayseri̇, Erciyes

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Tortella BJ, Carr ME, Rendo P, Korth-Bradley J, Smith LM, Kavakli K. Once-weekly prophylaxis regimen of nonacog alfa in patients with hemophilia B: an analysis of timing of bleeding event onset. Blood Coagul Fibrinolysis. 2021 Apr 1;32(3):180-185. doi: 10.1097/MBC.0000000000001012. PMID 33631774
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1821010&StudyName=Study%20To%20Compare%20On-Demand%20Treatment%20To%20A%20Prophylaxis%20Regimen%20Of%20BeneFIX%20In%20Subjects%20With%20Moderately%20Severe%20to%20Severe%20Hemophilia%20B

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participation included 25 enrolled participants from 15 study centers and 9 countries.
Pre-assignment Details: The duration of participation was approximately 86 weeks, consisting of a Screening period (1 day to 4 weeks), Period 1 (on-demand treatment for 26 weeks), Period 2 (prophylaxis therapy for 52 weeks), and a follow-up safety period (4 weeks).
Groups:
- All Participants: The data for all the participants is presented.
Period: Overall Study
Arm/Group | All Participants
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31.3 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Annualized Number of Bleeding Episodes.
Description: The annualized bleed rate (ABR) or the annualized number of bleeding episodes per year, will be derived for each participant for each treatment period by using the following formula: ABR = number of bleeds / (Days on treatment period / 365.25) The number of bleeds for the ABR calculation includes all bleeds requiring treatment with factor IX product during the time on treatment.
Time Frame: 2 years
Population: The efficacy analysis set (EAS) was used for the primary efficacy analyses with respect to ABR. It includes all participants who participated in at least one day of the routine prophylaxis period (ie, in the study through at least Visit 4).
Measure: Mean (Standard Deviation); unit: Number of bleeds per year
Groups:
- On-Demand Therapy: Participants were treated for the bleeding events at the discretion of the study physician according to BeneFIX label.
- Prophylaxis Therapy: The prophylaxis regimen of approximately 100 IU/kg once weekly was initiated at Visit 4.
Arm/Group | On-Demand Therapy | Prophylaxis Therapy
Number analyzed (Participants) | 25 | 25
Number of bleeds per year | 32.9 (17.4) | 3.6 (4.6)
Statistical Analysis 1: Comparison: On-Demand Therapy vs Prophylaxis Therapy; Test type: Superiority or Other; p < 0.0001, Paired t-test

2. Secondary Outcome: Response to On-Demand Treatment for All Bleeding Episodes.
Description: Assessment scores on a 4-point Response Scale for an on-demand bleeding episode, as assessed by participant/caregiver or investigator/qualified staff. The 4-point scale assessments are Excellent, Good, Moderate or No response. Responses to number of observations were noted.
Time Frame: 2 years
Population: The safety analysis set (SAS) was any participant who received at least one dose of BeneFIX, including the dose given during the enrollment visit (Visit 2) for the factor IX (FIX) recovery study. Follow-up infusion was only required for 18 participants.
Measure: Number; unit: Number of observations with response
Units Other Than Participants: bleeds
Groups:
- On-Demand Therapy-First Infusion; On-Demand Therapy-Follow-up Infusions: Participants were treated for the bleeding events at the discretion of the study physician according to BeneFIX label.
Arm/Group | On-Demand Therapy-First Infusion | On-Demand Therapy-Follow-up Infusions
Number analyzed (Participants) | 25 | 18
Number analyzed (bleeds) | 507 | 152
Number of observations with response
  Excellent | 271 | 39
  Good | 177 | 80
  Moderate | 55 | 33
  No response | 3 | 0
  Data not recorded | 1 | 0

3. Secondary Outcome: Number of Nonacog Alfa, Recombinant Factor IX (BeneFIX) Infusions Used to Treat Each Bleeding Episode.
Description: The number of study drug infusions administered to treat a bleed will be calculated by adding the initial (on-demand) infusion to any subsequent (on-demand) infusions for the same bleed (same bleed start date/time). The number of infusions needed to treat a bleed will be classified into the following categories: 1, 2, 3, 4 and >4 infusions. If there were more than one bleed location (e.g., ankle and joint) with identical bleed start date and time, it was treated as one bleed occurrence.
Time Frame: 2 years
Population: The safety analysis set (SAS) was any participant who received at least one dose of BeneFIX, including the dose given during the enrollment visit (Visit 2) for the factor IX (FIX) recovery study.
Measure: Number; unit: Number of bleeds requiring infusion
Units Other Than Participants: bleeds
Groups:
- All Population: The data for all the participants is presented.
Arm/Group | All Population
Number analyzed (Participants) | 25
Number analyzed (bleeds) | 507
Number of bleeds requiring infusion
  Number of Infusion: 1 | 416
  Number of Infusions: 2 | 69
  Number of Infusions: 3 | 9
  Number of Infusions: 4 | 3
  Number of Infusions: >4 | 10

4. Secondary Outcome: Number of Breakthrough (Spontaneous/Non-Traumatic) Bleeds Within 48 Hours of a Prophylaxis Dose of BeneFIX.
Description: The number of spontaneous, non-traumatic breakthrough bleeds within 48 hours following a prophylaxis dose of BeneFIX were summarized. If there was more than one bleed location (eg, ankle and joint) with identical bleed start date and time, it was treated as one bleed occurrence.
Time Frame: 2 years
Population: The safety analysis set (SAS) was any participant who received at least one dose of BeneFIX, including the dose given during the enrollment visit (Visit 2) for the factor IX (FIX) recovery study. Three participants experienced 1 spontaneous bleeding episode each within 48 hours of a previous prophylaxis infusion.
Measure: Mean (Standard Deviation); unit: Number of breakthrough bleeds
Units Other Than Participants: breakthrough bleeds
Arm/Group | All Participants
Number analyzed (Participants) | 25
Number analyzed (breakthrough bleeds) | 3
Number of breakthrough bleeds | 1.0 (0.0)

5. Secondary Outcome: Average Infusion Dose.
Description: The mean dose by per infusion by weight (IU/kg) was reported for both prophylaxis and on demand infusions
Time Frame: 2 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/Kg
Groups:
- Prophylaxis Therapy: The prophylaxis regimen of approximately 100IU/kg once weekly was initiated at Visit 4.
Arm/Group | On-Demand Therapy | Prophylaxis Therapy
Number analyzed (Participants) | 25 | 25
IU/Kg | 52 (16) [20 to 54] | 99 (2) [93 to 104]

6. Secondary Outcome: Total Factor Consumption.
Description: The total amount (IU) infused for each infusion recorded were summed to calculate the total factor consumption for each participant. For each infusion, IU/kg was calculated, using the most recently recorded weight measurement and the total factor consumption, divided by number of infusions, and was summarized similarly to average infusion dose (IU). Annualized TFC by weight was reported. Annualized TFC by weight = (Total IU/kg / treatment interval duration)*365.25.
Time Frame: 2 years
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: IU/Kg
Arm/Group | On-Demand Therapy | Prophylaxis Therapy
Number analyzed (Participants) | 25 | 25
IU/Kg | 707 (519) | 4985 (233)

7. Secondary Outcome: Incidence of Less Than Expected Therapeutic Effect (LETE)
Description: The following criteria are the definitions for LETE in this study: 1. LETE in the On-Demand Setting: LETE occurs in the on-demand setting if 2 successive "No Response" ratings are recorded after 2 successive BeneFIX drug infusions in the absence of confounding factors. 2. LETE in the Prophylaxis Setting: LETE occurs in the prophylaxis setting if there is a spontaneous bleed within 48 hours (≤ 48 hours) after a regularly scheduled prophylactic dose of BeneFIX in the absence of confounding factors. 3. LETE (Low Recovery): LETE can also be lower than expected recovery of FIX in the opinion of the investigator following infusion of BeneFIX in the absence of confounding factors. Each reported occurrence of low recovery LETE was listed.
Time Frame: 2 years
Population: as for outcome 3
Measure: Number; unit: Percentage of occurence
Arm/Group | All Participants
Number analyzed (Participants) | 25
Percentage of occurence
  LETE in On-Demand setting | 0
  LETE in prophylaxis setting | 0
  LETE (Low recovery) | 0

ADVERSE EVENTS:
Time Frame: Until follow-up 82 weeks +/- 4 days.
Description: Five participants experienced six SAEs since one participant experienced the same event twice (nephrolithiasis).
Arm/Group | On-Demand Therapy | Prophylaxis Therapy
Serious Adverse Events (participants affected / at risk) | 1/25 | 4/25
Other Adverse Events (participants affected / at risk) | 16/25 | 20/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | On-Demand Therapy (N=25) | Prophylaxis Therapy (N=25)
Pain (General disorders) | 0 | 1
Varicella (Infections and infestations) | 0 | 1
Blood pressure decreased (Investigations) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | On-Demand Therapy (N=25) | Prophylaxis Therapy (N=25)
Upper respiratory tract infection (Infections and infestations) | 4 | 5
Pharyngitis (Infections and infestations) | 2 | 3
Nasopharyngitis (Infections and infestations) | 3 | 1
Influenza (Infections and infestations) | 2 | 1
Inappropriate schedule of drug administration (Injury, poisoning and procedural complications) | 0 | 6
Drug dose omission (Injury, poisoning and procedural complications) | 0 | 4
Medication error (Injury, poisoning and procedural complications) | 0 | 3
Underdose (Injury, poisoning and procedural complications) | 0 | 3
Wrong dose administration (Injury, poisoning and procedural complications) | 0 | 3
Head injury (Injury, poisoning and procedural complications) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 8 | 4
Toothache (Gastrointestinal disorders) | 3 | 5
Gastritis (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Pyrexia (General disorders) | 4 | 4
Local swelling (General disorders) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.